CLINICAL TRIAL: NCT03551171
Title: An Open-Label,Single-Arm,Phase I Clinical Trial to Evaluate the Pharmacokinetics,Safety and Tolerability of ZL-2306 (Niraparib) in Patients With Ovarian Cancer,Fallopian Tube Cancer and Primary Peritoneal Cancer (Collectively Termed as Ovarian Cancer)
Brief Title: The Clinical Trial to Evaluate the Pharmacokinetics, Safety and Tolerability of ZL-2306 (Niraparib) in Patients With Ovarian Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zai Lab (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Zai Lab (Hong Kong), Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZL-2306-002
Record Dates: First submitted 2018-04-20; First posted 2018-06-11 (Actual); Last update posted 2019-01-24 (Actual); Status verified 2018-05

CONDITIONS: Ovarian Cancer
Keywords: PARP inhibitor; BRCA mutation
MeSH Terms: conditions — Ovarian Neoplasms | interventions — niraparib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ZL-2306 (niraparib) (Experimental): Subjects will be randomised into 100mg, 200mg, 300mg dose group at the first day of the first cycle.
  Interventions: Drug: ZL-2306 (niraparib)

INTERVENTIONS:
Drug: ZL-2306 (niraparib) — About 30 subjects will be enrolled to the study, and randomised into 300mg, 200mg and 100mg dose groups (about 10 subjects per group).
  All subjects will be randomised into indicated dose group (300mg, 200mg or 100mg) at the first day of the first cycle. A single administration of ZL-2306 (niraparib) will be given to the subjects at indicated dose.

SUMMARY:
Niraparib is a potent and highly selective PARP-1/-2 inhibitor. The primary objective of this trial is to evaluate the pharmacokinetic (PK) properties of ZL-2306 (niraparib) and its metabolite M1 in patients from Mainland China with ovarian cancer, following a single and multiple oral administration of the study drug at the indicated dose (300mg, 200mg or 100mg), once a day.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent .
2. Female, age ≥ 18 years.
3. Histologically confirmed diagnosis of FIGO stage III or IV ovarian cancer, fallopian tube cancer, or primary peritoneal cancer.
4. Has received no further than second-line platinum-based chemotherapy, and has clinical complete response (CR) or partial response (PR) at least following 4 courses of the last platinum-based chemotherapy.
5. ECOG 0-1.
6. Has good organ function, including:
7. Patient of childbearing potential, has a negative pregnancy test when enrolled and promises to use an adequate method of contraception or abstain from activities that could result in pregnancy from enrolment to the end of study and during the 3 months after the last dose of the study treatment, or be of non-childbearing potential, can be enrolled in the study.
8. Is able to adhere to the protocol.
9. Has recovered from previous chemotherapy induced toxic side effects to ≤ grade 1 CTCAE or basal level, apart from ≤ grade 2 CTCAE peripheral neuropathy or hair loss symptoms at steady state.

Exclusion Criteria:

1. Has a known hypersensitivity to the active or inactive ingredients of ZL-2306 (niraparib) or compound which has similar chemical structure to ZL-2306 (niraparib).
2. Has symptomatic uncontrolled brain or leptomeningeal metastasis.
3. Major surgery or chemotherapy within 3 weeks of starting the study or patient has not recovered from any effects of the surgery.
4. Receive palliative radiotherapy encompassing > 20% of the bone marrow within 1 week of entering the study.
5. Be diagnosed any invasive cancer other than ovarian cancer (apart from cured basal cell carcinoma and squamous cell carcinoma) within 2 years prior to study enrolment.
6. Has a history or current diagnosis of myelodysplastic syndrome (MDS) and acute myeloid leukaemia (AML).
7. Has other serious or uncontrolled disease
8. Has any disease, treatment and laboratory abnormality that may interfere the study results and affect the fully attendance of study. Or the patient is considered to be not suitable for the study by the investigator. Cannot receive platelet or red blood cell transfusion within 4 weeks of study drug administration.
9. Pregnant, breastfeeding or expecting to conceive children during the study treatment period.
10. Corrected QT (QTc) interval > 470 msec.
11. Use proton pump inhibitors, antacids or histamine 2 (H2) blockers within 48hrs prior to the first drug administration for PK measurement.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2017-12-19 (Actual); Primary Completion 2018-05-03 (Actual); Study Completion 2018-07-10 (Actual)

PRIMARY OUTCOMES:
Maximum plasma drug concentration (Cmax) | From pre-dose to day 1 of the 2nd cycle (each cycle is 28 days)
Time to reach Cmax (Tmax) | From pre-dose to day 1 of the 2nd cycle (each cycle is 28 days)
Terminal rate constant (λz) | From pre-dose to day 1 of the 2nd cycle (each cycle is 28 days)
Elimination half-life (t1/2) | From pre-dose to day 1 of the 2nd cycle (each cycle is 28 days)
Area under the plasma concentration-time curve from time zero to 24hrs (AUC (0-24)) | From pre-dose to day 1 of the 2nd cycle (each cycle is 28 days)
Area under the plasma concentration-time curve from time zero to time of last measurable concentration (AUC(0-t)) and from zero to infinity (AUC0-∞) | From pre-dose to day 1 of the 2nd cycle (each cycle is 28 days)
Apparent total body clearance of the drug from plasma (CL/F) | From pre-dose to day 1 of the 2nd cycle (each cycle is 28 days)
Apparent volume of distribution (Vd/f) | From pre-dose to day 1 of the 2nd cycle (each cycle is 28 days)
Mean residence time (MRT) | From pre-dose to day 1 of the 2nd cycle (each cycle is 28 days)
Degree of fluctuation (DF) | From pre-dose to day 1 of the 2nd cycle (each cycle is 28 days)
Maximum plasma drug concentration at steady-state (Css max) | From pre-dose to day 1 of the 2nd cycle (each cycle is 28 days)
Time to reach Css max (Tss max) | From pre-dose to day 1 of the 2nd cycle (each cycle is 28 days)
Minimum plasma drug concentration at steady-state (Css min) | From pre-dose to day 1 of the 2nd cycle (each cycle is 28 days)
Area under the plasma concentration-time curve from time zero to the end of drug administration (AUCss) | From pre-dose to day 1 of the 2nd cycle (each cycle is 28 days)
Steady-state apparent total body clearance of drug from plasma (Clss/F) | From pre-dose to day 1 of the 2nd cycle (each cycle is 28 days)
Accumulation ratio following multiple drug administration (RAC) | From pre-dose to day 1 of the 2nd cycle (each cycle is 28 days)
The plasma drug concentration before drug administration | From pre-dose to day 1 of the 2nd cycle (each cycle is 28 days)

SECONDARY OUTCOMES:
Number of participants with adverse events as assessed by CTCAE v4.0 | From the signing of ICF till the end of this study (30 days after the last administration of the study drug or the date to close the clinical trial database, whichever is earlier)

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Haerbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Hunan Cancer Hospital, Changsha, Hunan
  - Fudan University Shanghai Cnacer Center, Shanghai, Shanghai Municipality
  - The West China Second UniversityHospital of Sichuan University, Chengdu, Sichuan

REFERENCES:
- [Derived] Zhang J, Zheng H, Gao Y, Lou G, Yin R, Ji D, Li W, Wang W, Xia B, Wang D, Hou J, Yan J, Hei Y, Zhang ZY, Milton A, Wu X. Phase I Pharmacokinetic Study of Niraparib in Chinese Patients with Epithelial Ovarian Cancer. Oncologist. 2020 Jan;25(1):19-e10. doi: 10.1634/theoncologist.2019-0565. Epub 2019 Aug 22. PMID 31439812